CLINICAL TRIAL: NCT02022605
Title: Effect of Continuously Coached Practice Using EMS on ERCP Performance of Trainees: a Prospectively Randomized, Controlled Study
Brief Title: Effect of Continuously Coached Practice Using EMS on ERCP Performance of Trainees
Acronym: ERCP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 20131208-4; 20131208-4 (Other: Ethics committee of Xijing Hospital)
Record Dates: First submitted 2013-12-21; First posted 2013-12-30 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Selective Cannulation Rate of Trainees Receiving ERCP Training
Keywords: ERCP, trainning, trainees, EMS

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hands-on EMS training group (Experimental)
  Interventions: Device: Hands-on EMS training; Other: Standard training
- Standard training group (Active Comparator)
  Interventions: Other: Standard training

INTERVENTIONS:
Device: Hands-on EMS training — A trainer (SAH) gave a series of demonstrations of the proper techniques of ERCP step by step on the EMS. The demonstration included selective cannulation, sphincterotomy, guidewire exchange, balloon dilation, stone extraction and stent insertion. Then trainees practiced each technique with hands-on coaching from the trainer on the EMS. Each trainee could repeate the practice with the trainer giving only verbal correction of any errors for about 30min.
  Arms: Hands-on EMS training group
Other: Standard training — The standard cannulation technique was used with a sphincterotome preloaded with a guidewire, positioned in the ampullary orifice, and targeting the presumed entry of CBD or PD. During the whole procedure of cannulation by trainees, the senior endoscopist would actively communicate with trainees through verbal and/or hands-on assistance to help them to make the performance more correctly. If the trainees failed to enter the targeted duct within 10min, the senior endoscopist would take over the duodenoscope and continue the following procedure of cannulation.

SUMMARY:
Previous studies have demonstrated that coached EMS practice at the beginning of ERCP training could improve the trainees' skill. However, it is not known whether continuously coached practice using EMS can provide additional benefit.

ELIGIBILITY:
Inclusion Criteria:

* consecutive inpatients with naive papilla undergoing ERCP.

Exclusion Criteria:

* history of partial or total gastrectomy (Billroth I/II, Roux-en-Y);
* duodenal stricture (benign or melignant);
* ampullary carcinoma;
* previously failed selective cannulation;
* chronic pancreatitis with PD stone;
* minor papilla cannulation;
* servere diseases of heart, lung, brain and kidney;
* hemodynamical unstablility;
* pregnant women;
* refusal or unable to give written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of selective cannulation in 10min by trainee | 2 years

SECONDARY OUTCOMES:
Total time of successful cannulation | 2 years
Cumulative success rate of each month | 2 years
Performance score of selective cannulation | 2 years
Performance score of EST | 2 years
Complication rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, M.D., Principal Investigator — Xijing Hospital of Digestive Diseases.The Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Liao WC, Leung JW, Wang HP, Chang WH, Chu CH, Lin JT, Wilson RE, Lim BS, Leung FW. Coached practice using ERCP mechanical simulator improves trainees' ERCP performance: a randomized controlled trial. Endoscopy. 2013 Oct;45(10):799-805. doi: 10.1055/s-0033-1344224. Epub 2013 Jul 29. PMID 23897401
- [Background] Lim BS, Leung JW, Lee J, Yen D, Beckett L, Tancredi D, Leung FW. Effect of ERCP mechanical simulator (EMS) practice on trainees' ERCP performance in the early learning period: US multicenter randomized controlled trial. Am J Gastroenterol. 2011 Feb;106(2):300-6. doi: 10.1038/ajg.2010.411. Epub 2010 Oct 26. PMID 20978485